CLINICAL TRIAL: NCT02253160
Title: A Randomized, Crossover Trial to Characterize the Performance of the Spectra Optia Apheresis System Versus the COBE Spectra Apheresis System for Collection of Mononuclear Cells in Healthy Adult Donors
Brief Title: An Evaluation of the Spectra Optia CMNC Collection Procedure
Acronym: CMNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CTS-5038
Record Dates: First submitted 2014-09-23; First posted 2014-10-01 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Apheresis Donors; Mononuclear (MNC) Cell Donors
Keywords: MNCs; Mononuclear Cells; Apheresis; Spectra Optia
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spectra Optia CMNC first, then COBE Spectra MNC (Experimental): Spectra Optia CMNC collection procedure followed by COBE Spectra MNC collection procedure.
  Interventions: Device: Spectra Optia CMNC; Device: COBE Spectra MNC; Drug: Granulocyte-colony stimulating factor (G-CSF)
- COBE Spectra MNC first, then Spectra Optia CMNC (Experimental): COBE Spectra MNC collection procedure followed by Spectra Optia CMNC collection procedure.
  Interventions: Device: Spectra Optia CMNC; Device: COBE Spectra MNC; Drug: Granulocyte-colony stimulating factor (G-CSF)

INTERVENTIONS:
Device: Spectra Optia CMNC — The Spectra Optia® Apheresis System is an automated centrifugal system that separates whole blood into its cellular and plasma components. The device is comprised of three major sub-systems, 1) the apheresis machine itself (centrifuge, centrifuge filler, pumps, valves, computerized safety and control systems, etc.), 2) a sterile, single-use, disposable blood tubing set, and 3) embedded software. The Spectra Optia system's investigational CMNC procedure will be used to collect MNC from the peripheral blood.
  Other Names: Spectra Optia Apheresis System CMNC collection procedure
Device: COBE Spectra MNC — It is also a centrifugal system that separates whole blood into its cellular and plasma components. The COBE Spectra MNC collection procedure is chosen as the comparator device because it is the reference after which design of the Spectra Optia CMNC collection procedure was modeled.
  Other Names: COBE Spectra Apheresis System MNC collection procedure
Drug: Granulocyte-colony stimulating factor (G-CSF) — Each subject received an injection of the G-CSF approximately equivalent to 10 ug/kg body weight subcutaneous per day for 5 days prior to the MNC collection procedure.
  Other Names: Mobilization Procedure

SUMMARY:
The purpose of this prospective, randomized, cross-over, multi-center study is to evaluate the performance of the Spectra Optia Apheresis System's CMNC Collection Procedure, compared to the COBE Spectra Apheresis System's MNC Procedure in mobilized healthy donors. Subject safety will be evaluated beginning with mobilization, throughout the collection procedure and for the day following the last collection.

DETAILED DESCRIPTION:
This is a prospective, randomized, cross-over, multi-center study to evaluate the performance of the Spectra Optia system's CMNC Collection Procedure, compared to the COBE Spectra system's MNC Procedure in mobilized healthy donors.

Up to 60 subject may be consented to meet the the enrollment target of 20 complete subjects. Eligible subjects will be randomized to receive either the Spectra Optia CMNC or the COBE Spectra MNC collection procedure first, followed by the opposite on the following day.

Study participation will be up to 14 days: a 7-day screening period, four days for mobilization, one day for the first MNC collection with additional dose of mobilization, one day for the second MNC collection, and safety follow-up the following day.

Subject safety will be evaluated beginning with mobilization, throughout the collection procedure and for the day following the second collection.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 and ≤ 50 years of age
2. Healthy blood donor criteria as defined by the American Associate of Blood Banks (AABB)

   a) Note: Subjects who are deferred from volunteer donations because of travel restrictions, piercings or tattoos may participate in the study
3. Adequate dual peripheral venous access
4. Acceptable prescreening laboratory results prior to MNC mobilization as specified below:

   a) WBC 3,500 - 10,800/µL

   b) Hematocrit 38% - 56%

   c) Platelets 150,000 - 400,000/µL

   d) Coagulation tests:

   i. PT 9.0 - 13.0 seconds

   ii. PTT 23.4 - 41.8 seconds

   e) Serum electrolytes:

   i. Potassium 3.6 - 5.1 mmol/L

   ii. Serum Calcium 8.5 mg/dL - 10.3 mg/dL

   f) Renal function: Serum creatinine ≤ 1.5 mg/dL

   NOTE: up to two laboratory results may fall out of the ranges listed above if, in the judgment of the investigator, they do not constitute a significant risk to the subject.
5. Liver function: alanine aminotransferase (ALT) < 1.5 times the upper limit of normal
6. Willing to avoid pregnancy until at least 48 hours following last G-CSF injection

   1. If male, be willing to use a condom during sexual relations with a female partner until 48 hours following the last G-CSF injection
   2. If female and of childbearing potential, be willing to use a medically acceptable contraceptive until 48 hours following the last G-CSF injection
7. Given written informed consent

Exclusion Criteria:

1. Previous MNC collection failure
2. Known hypersensitivity or condition that prevents the use of anticoagulants
3. Known hypersensitivity or condition that prevents the use of G-CSF
4. Known hemoglobinopathy including sickle cell trait or disease
5. History of use in the past week or anticipated need for lithium
6. Concurrent enrollment in another clinical study that could impact the results or participation in this study
7. Active infection or any serious underlying medical condition that contraindicates apheresis
8. Women who are pregnant or lactating
9. Known history of significant head trauma

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Goodrich, PhD, Study Director — Terumo BCT
Locations (2):
- United States (2):
  - Hoxworth Blood Center, Cincinnati, Ohio
  - Key Biologics, LLC, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the specialized donor population of blood centers from August 2014 through January 2015.
Pre-assignment Details: A lead-in phase was used to allow for investigational device training. One subject consented the lead-in phase and was included in the safety analysis only. After a screening period to evaluate and confirm eligibility criteria prior to enrollment & randomization to treatment assignment (Arm 1 or Arm 2) 22 subjects enrolled in the pivotal study.
Groups:
- Lead-in Donor: Subjects screened and enrolled for the purpose of training on the investigational procedure only. Included in safety analysis only.
Period: Overall Study
Arm/Group | Lead-in Donor | Spectra Optia CMNC First, Then COBE Spectra MNC | COBE Spectra MNC First, Then Spectra Optia CMNC
Started | 1 | 12 | 10
Completed | 1 | 12 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Healthy adult specialized blood donors
Groups:
- Total: Total of all reporting groups
Arm/Group | Lead-in Donor | Spectra Optia CMNC First, Then COBE Spectra MNC | COBE Spectra MNC First, Then Spectra Optia CMNC | Total
Number analyzed (Participants) | 1 | 12 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (NA) — no s.d. available when n=1 | 35.4 (7.32) | 34.8 (8.44) | 35.0 (7.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 3
  Male | 1 | 11 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 12 | 10 | 23
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 6 | 12
  White | 0 | 6 | 4 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Weight [Mean (Standard Deviation); unit: kilograms] | 110 (NA) — no s.d. available when n=1 | 115.23 (28.921) | 97.08 (26.654) | 107.11 (28.124)
Height [Mean (Standard Deviation); unit: inches] | 60 (NA) — no s.d. available when n=1 | 70.8 (2.45) | 69.4 (4.06) | 69.7 (3.83)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 47.36 (NA) — no s.d. available when n=1 | 35.82 (9.413) | 30.88 (6.050) | 34.17 (8.579)

OUTCOME MEASURES:

1. Primary Outcome: CD34+ Collection Efficiency (CE1 %)
Description: The primary endpoint is the CD34+ cell collection efficiency (CE) associated with the Mononuclear Cell (CMNC) Collection Procedures on the Spectra Optia and COBE Spectra Apheresis Systems. CE is a measurement of device performance calculated using donor and blood product blood counts collected immediately before and after the CMNC collection procedure. The collection efficiency for a given cell type is defined as the percent of processed cells of that cell type that are in fact collected.
Time Frame: within 5 minutes upon completion of procedure
Measure: Mean (Standard Deviation); unit: percent
Groups:
- Treatment Assignment 1: Spectra Optia CMNC collection procedure followed by COBE Spectra MNC collection procedure.
  Spectra Optia CMNC: The Spectra Optia® Apheresis System is an automated centrifugal system that separates whole blood into its cellular and plasma components. The device is comprised of three major sub-systems, 1) the apheresis machine itself (centrifuge, centrifuge filler, pumps, valves, computerized safety and control systems, etc.), 2) a sterile, single-use, disposable blood tubing set, and 3) embedded software. The Spectra Optia system's investigational CMNC procedure will be used to collect MNC from the peripheral blood.
  COBE Spectra MNC: It is also a centrifugal system that separates whole blood into its cellular and plasma components. The COBE Spectra MNC collection procedure is chosen as the comparator device because it is the reference after which design of the Spectra Optia CMNC collection procedure was modeled.
- Treatment Assignment 2: COBE Spectra MNC collection procedure followed by Spectra Optia CMNC collection procedure.
  Spectra Optia CMNC: The Spectra Optia® Apheresis System is an automated centrifugal system that separates whole blood into its cellular and plasma components. The device is comprised of three major sub-systems, 1) the apheresis machine itself (centrifuge, centrifuge filler, pumps, valves, computerized safety and control systems, etc.), 2) a sterile, single-use, disposable blood tubing set, and 3) embedded software. The Spectra Optia system's investigational CMNC procedure will be used to collect MNC from the peripheral blood.
  COBE Spectra MNC: It is also a centrifugal system that separates whole blood into its cellular and plasma components. The COBE Spectra MNC collection procedure is chosen as the comparator device because it is the reference after which design of the Spectra Optia CMNC collection procedure was modeled.
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 12 | 10
percent
  Spectra Optia | 87.7 (20.18) | 81.4 (10.24)
  COBE Spectra | 66.6 (20.26) | 65.8 (6.40)

2. Secondary Outcome: CD34+ Collection Efficiency (CE2 %)
Description: Comparison of collection efficiencies associated with the CMNC Cell Collection Procedures on the Spectra Optia and COBE Spectra Apheresis Systems. CE is a measurement of device performance calculated using donor blood counts immediately before and blood product blood counts immediately after the collection procedure. The collection efficiency for a given cell type is defined as the percent of processed cells of that cell type that are in fact collected.
Time Frame: within 5 minutes upon completion of procedure
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 12 | 10
percent
  Spectra Optia | 64.7 (14.61) | 59.6 (6.17)
  COBE Spectra | 47.0 (14.86) | 50.2 (4.20)

3. Secondary Outcome: MNC Collection Efficiency (CE1%)
Description: Comparison of collection efficiencies associated with the CMNC Collection Procedures on the Spectra Optia and COBE Spectra Apheresis Systems for MNCs. CE1 is a measurement of device performance calculated using donor and blood product blood counts collected immediately before and after the collection procedure. The collection efficiency for a given cell type is defined as the percent of processed cells of that cell type that are in fact collected.
Time Frame: within 5 minutes upon completion of procedure
Population: One subject was not included in MNC CE1 because of missing MNC lab results post-collection, therefore CE1 could not be calculated.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 11 | 10
percent
  Spectra Optia CE1 | 62.06 (17.220) | 63.75 (18.900)
  COBE Spectra CE1 | 45.46 (6.483) | 48.58 (14.685)

4. Secondary Outcome: CD34+ Per kg of Body Weight
Time Frame: within 5 minutes upon completion of procedure
Measure: Mean (Standard Deviation); unit: cells/kg
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 12 | 10
cells/kg
  Spectra Optia | 5.14 (3.756) | 3.75 (1.506)
  COBE Spectra | 3.50 (2.732) | 3.68 (1.546)

5. Secondary Outcome: MNC Product Contamination/Purity (%) - Hematocrit (%)
Time Frame: within 5 minutes upon completion of procedure
Measure: Mean (Standard Deviation); unit: % of red blood cells
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 12 | 10
% of red blood cells
  Spectra Optia Hematocrit | 6.1 (2.12) | 3.7 (0.95)
  COBE Spectra Hematocrit | 4.5 (1.54) | 5.7 (1.71)

6. Secondary Outcome: MNC Product Contamination/Purity (%) - Granulocyte Concentration (10^3/mL)
Time Frame: within 5 minutes upon completion of procedure
Measure: Mean (Standard Deviation); unit: cells*10^3/mL
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 12 | 10
cells*10^3/mL
  Spectra Optia | 51.689 (35.5970) | 63.338 (44.9682)
  COBE Spectra | 83.792 (58.9491) | 70.944 (72.4223)

7. Secondary Outcome: MNC Product Contamination/Purity (%) - Platelet Concentration (10^3/µL)
Time Frame: within 5 minutes upon completion of procedure
Measure: Mean (Standard Deviation); unit: cells*10^3/µL
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 12 | 10
cells*10^3/µL
  Spectra Optia | 3724.9 (962.42) | 2022.9 (674.91)
  COBE Spectra | 2857.4 (467.44) | 3736.0 (1200.88)

8. Secondary Outcome: MNC Product Contamination/Purity (%) - Platelet Collection Efficiency (CE1 %)
Description: Comparison of collection efficiencies associated with the CMNC Collection Procedures on the Spectra Optia and COBE Spectra Apheresis Systems for platelets. CE1 is a measurement of device performance calculated using donor and blood product blood counts collected immediately before and after the collection procedure. The collection efficiency for a given cell type is defined as the percent of processed cells of that cell type that are in fact collected.
Time Frame: within 5 minutes upon completion of procedure
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 11 | 10
percent
  Spectra Optia | 28.7 (14.08) | 23.5 (8.62)
  COBE Spectra | 27.9 (9.19) | 30.3 (9.85)

9. Secondary Outcome: MNC Blood Product Volume (mL)
Description: The produced unit of MNCs collected into the blood bag.
Time Frame: within 5 minutes upon completion of procedure
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 12 | 10
mL
  Spectra Optia | 144.8 (32.99) | 141.3 (30.82)
  COBE Spectra | 140.8 (28.36) | 137.7 (28.64)

10. Secondary Outcome: Purity of Plasma Collected for Laboratory Processing of MNC Product - Platelet Concentration in Plasma (10^3/µL)
Description: A small amount of plasma typically used for processing was collected in a sub-set of collection procedures.
Time Frame: within 5 minutes upon completion of procedure
Population: Five collections also collected plasma for this sub-study.
Measure: Mean (Standard Deviation); unit: cells*10^3/µL
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 2 | 3
cells*10^3/µL
  Spectra Optia | 32.5 (30.41) | 8.7 (5.86)
  COBE Spectra | 147.5 (4.95) | 179.3 (72.47)

11. Secondary Outcome: Procedure Time (Minutes)
Time Frame: within 5 minutes upon completion of procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 12 | 10
minutes
  Spectra Optia | 153.8 (30.90) | 151.4 (27.55)
  COBE Spectra | 151.1 (31.92) | 146.7 (27.35)

12. Other Pre Specified Outcome: Device Deficiencies
Description: Any time a device or disposable does not function as described in the Operator's Manual or Package Insert, a Device Deficiency must be reported. This includes those instances wherein Operator Error led to a malfunction/deficiency. A device deficiency is any inadequacy in the identity, quality, durability, reliability, safety or performance of an investigational device, including malfunction, use errors or inadequacy in the information supplied by the manufacturer. Device malfunctions and device incidents should be reported in the same manner.
Time Frame: 24-hours after last collection procedure
Population: All pivotal subjects (n=22) received both the Spectra Optia and the COBE Spectra per the crossover design. The lead-in subject only received the Spectra Optia. Both lead-in and pivotal subjects are included in any safety analysis.
Measure: Number; unit: events
Groups:
- Spectra Optia: Subjects who received an CMNC collection using the Spectra Optia
- COBE Spectra: Subjects who received an CMNC collection using the COBE Spectra
Arm/Group | Spectra Optia | COBE Spectra
Number analyzed (Participants) | 23 | 22
events | 1 | 0

13. Other Pre Specified Outcome: Post-collection Platelet Loss in Subject
Description: The percent change from pre-collection platelet count to post-collection subject platelet count.
Time Frame: 24-hours after last collection procedure
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 12 | 10
percent change
  Spectra Optia | 27.2 (9.88) | 23.9 (8.04)
  COBE Spectra | 27.2 (9.42) | 30.7 (6.18)

14. Secondary Outcome: MNC Collection Efficiency (CE2%)
Description: Comparison of collection efficiencies associated with the CMNC Collection Procedures on the Spectra Optia and COBE Spectra Apheresis Systems for MNCs. CE2 is a measurement of device performance calculated using donor blood counts immediately before and blood product counts immediately after the collection procedure and does not average the donor pre- and post-collection counts. The collection efficiency for a given cell type is defined as the percent of processed cells of that cell type that are in fact collected.
Time Frame: within 5 minutes upon completion of procedure
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 12 | 10
percent
  Spectra Optia CE2 | 50.99 (16.590) | 52.98 (17.528)
  COBE Spectra CE2 | 37.77 (5.297) | 39.72 (13.972)

15. Secondary Outcome: MNC Product Contamination/Purity - RBC Concentration (10^6/µL)
Time Frame: within 5 minutes upon completion of procedure
Measure: Mean (Standard Deviation); unit: RBC*10^6/µL
Arm/Group | Treatment Assignment 1 | Treatment Assignment 2
Number analyzed (Participants) | 12 | 10
RBC*10^6/µL
  Spectra Optia RBC Concentration | 1.029 (0.4740) | 0.526 (0.1990)
  COBE Spectra RBC Concentration | 0.653 (0.2786) | 0.857 (0.2501)

ADVERSE EVENTS:
Time Frame: AEs were captured per protocol from the first dose of G-CSF until final follow up, which was typically 1 day after the last CMNC Collection Procedure for a total of 7 days.
Groups:
- Pre-collection: Subjects screened and received G-CSF.
- Spectra Optia: Subject who received Spectra Optia CMNC collection procedure.
- COBE Spectra: Subjects who received COBE Spectra MNC collection procedure.
- Follow up: Subjects who completed cross-over design and were followed for at least 1 day.
Arm/Group | Pre-collection | Spectra Optia | COBE Spectra | Follow up
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 22/23 | 13/23 | 16/22 | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-collection (N=23) | Spectra Optia (N=23) | COBE Spectra (N=22) | Follow up (N=23)
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 5 | 5 | 1
fatigue (General disorders) | 5 | 1 | 0 | 1
hemoglobin decreased (Investigations) | 2 | 3 | 2 | 0
platelet count decreased (Investigations) | 0 | 0 | 5 | 0
back pain (Musculoskeletal and connective tissue disorders) | 10 | 1 | 0 | 0
bone pain (Musculoskeletal and connective tissue disorders) | 9 | 0 | 0 | 0
paraesthesia (Nervous system disorders) | 1 | 1 | 2 | 0
palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 1 | 0
abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
infusion site extravasation (General disorders) | 0 | 1 | 0 | 0
injection site pain (General disorders) | 1 | 0 | 0 | 0
decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
musculoskeletal pain (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
headache (Nervous system disorders) | 0 | 0 | 1 | 0
neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 2
tension headach (Nervous system disorders) | 0 | 1 | 0 | 0
insomina (Psychiatric disorders) | 1 | 1 | 0 | 0
restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less